CLINICAL TRIAL: NCT04279821
Title: Prevalence of Segmental Colitis Associated With Colic Diverticulosis (SCAD): an Observational Study
Brief Title: Prevalence of Segmental Colitis Associated With Colic Diverticulosis (SCAD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Bruno Annibale, Full Professor, University of Roma La Sapienza
Other Study IDs: 263 SA_2019
Record Dates: First submitted 2020-02-13; First posted 2020-02-21 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Diverticular Disease of Colon; Diverticulosis, Colonic
Keywords: Segmental colitis associated with colic diverticulosis
MeSH Terms: conditions — Diverticulosis, Colonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colonic diverticulosis and macroscopic signs of inflammation: No interventional study

SUMMARY:
Colonic diverticula are common in Western countries, affecting up to 60% of subjects over 70 years of age. In about 80% of patients, colonic diverticula remain asymptomatic (diverticulosis), while approximately 20% of patients may develop abdominal symptoms (symptomatic uncomplicated diverticular disease, SUDD) and, eventually, complications such as bouts of diverticulitis or bleeding.

A small proportion of patients with colonic diverticulosis may develop segmental colitis associated with diverticulosis (SCAD). SCAD is separate clinical disease with specific macroscopic (erythema, friability and ulcerations) and microscopic features characterized by chronic, mucosal inflammation involving the inter-diverticular mucosa (usually sigmoid colon) sparing the proximal colon and rectum colon.

The most common symptoms of SCAD are rectal bleeding, diarrhoea and abdominal pain.

To achieve SCAD diagnosis a correct biopsies sampling is mandatory. It is necessary to take biopsies on the borders of the diverticula and in the apparently normal adjacent mucosa as well as biopsies in both the colon proximal to the diverticular area and the rectum in order to exclude chronic inflammatory bowel disease. The spectrum of histological lesions associated with SCAD is variable, including mild non-specific inflammation and inflammatory bowel disease (IBD)-like changes.

Currently, data regarding prevalence of SCAD are scarce. It has been estimated that in patients with diverticulosis, SCAD prevalence ranged from 0.3-1.3%.

The aim of the present study is to assess prospectively the prevalence of segmental colitis associated with colon diverticulosis (SCAD), in consecutive patients with colic diverticulosis, in a tertiary university centre.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic finding of colonic diverticulosis associated with macroscopic signs of inflammation (erythema, friability and ulcerations) of the interdiverticular mucosa

Exclusion Criteria:

* inability to sign informed consent;
* impossibility to perform biopsies during colonoscopy (e.g. anticoagulant therapy/ conditions predisposing to high risk of bleeding);
* Diagnosis of chronic inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients (>18 years of age) who perform a colonoscopy (for screening or other clinical/diagnostic reasons) during which diverticulosis of the colon is associated with macroscopic signs of inflammation (erythema, friability and ulcerations) of the interdiverticular mucosa, in a tertiary university centre.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Segmental Colitis Associated With Colic Diverticulosis (SCAD) as assessed by histology | 1 year
  Number of patients with histological diagnosis of SCAD in patients with endoscopic signs of inflammation of the interdiverticular mucosa

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Annibale, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- University Hospital Sant'Andrea, University Sapienza Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parra-Blanco A. Colonic diverticular disease: pathophysiology and clinical picture. Digestion. 2006;73 Suppl 1:47-57. doi: 10.1159/000089779. Epub 2006 Feb 8. PMID 16498252
- [Background] Stollman N, Raskin JB. Diverticular disease of the colon. Lancet. 2004 Feb 21;363(9409):631-9. doi: 10.1016/S0140-6736(04)15597-9. PMID 14987890
- [Background] Cuomo R, Barbara G, Pace F, Annese V, Bassotti G, Binda GA, Casetti T, Colecchia A, Festi D, Fiocca R, Laghi A, Maconi G, Nascimbeni R, Scarpignato C, Villanacci V, Annibale B. Italian consensus conference for colonic diverticulosis and diverticular disease. United European Gastroenterol J. 2014 Oct;2(5):413-42. doi: 10.1177/2050640614547068. PMID 25360320
- [Background] Freeman HJ. Natural history and long-term clinical behavior of segmental colitis associated with diverticulosis (SCAD syndrome). Dig Dis Sci. 2008 Sep;53(9):2452-7. doi: 10.1007/s10620-007-0173-y. Epub 2008 Mar 13. PMID 18338265